CLINICAL TRIAL: NCT02662335
Title: Computerized Cognitive Retraining in Breast Cancer Survivors
Brief Title: Computerized Cognitive Retraining in Improving Cognitive Function in Breast Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 9363; NCI-2015-02193 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 9363 (Other: Fred Hutch/University of Washington Cancer Consortium); P30CA015704 (NIH)
Record Dates: First submitted 2016-01-20; First posted 2016-01-25 (Estimated); Last update posted 2017-12-13 (Actual); Status verified 2017-12

CONDITIONS: Cancer Survivor; Stage 0 Breast Cancer; Stage IA Breast Cancer; Stage IB Breast Cancer; Stage IIA Breast Cancer; Stage IIB Breast Cancer; Stage IIIA Breast Cancer; Stage IIIB Breast Cancer; Stage IIIC Breast Cancer
MeSH Terms: conditions — Breast Carcinoma In Situ; Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (computer-assisted cognitive training) (Experimental): Patients complete a computerized working memory training program (Cogmed) over 35 minutes a day, 5 times a week for 6 weeks.
  Interventions: Other: Computer-Assisted Cognitive Training; Other: Questionnaire Administration
- Arm II (wait-list) (Active Comparator): Patients undergo standard follow-up care for 6 weeks. Following standard follow-up care, patients may complete Cogmed as in the Intervention Group in weeks 7-13.
  Interventions: Other: Questionnaire Administration; Procedure: Standard Follow-Up Care

INTERVENTIONS:
Other: Computer-Assisted Cognitive Training — Participate in Cogmed computerized working memory training
  Arms: Arm I (computer-assisted cognitive training)
Other: Questionnaire Administration — Ancillary studies
Procedure: Standard Follow-Up Care — Undergo standard follow-up care
  Arms: Arm II (wait-list)

SUMMARY:
This randomized clinical trial studies computerized cognitive retraining in improving cognitive function in breast cancer survivors. Cancer-related cognitive deficits, such as thinking and memory issues, are common among breast cancer survivors. The severity of these cognitive deficits is associated with a significant negative impact on daily function and quality of life. A computerized cognitive retraining method may help researchers find ways to improve cognitive function and quality of life in breast cancer survivors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Evaluate the feasibility and acceptability of a 6-week computerized working memory training program in breast cancer survivors who subjectively report cognitive deficits: evaluate feasibility of study procedures (recruitment and screening procedures, number of participants recruited, screened, and retained, attrition rate and reason, weekly phone calls completed with participants); evaluate the acceptability of an adaptive computerized working memory training intervention (burden, adherence to training schedule, performance level achieved, and participant satisfaction with computerized exercises).

SECONDARY OBJECTIVES:

I. To evaluate the difference in the posttest means at T2 (week #7) adjusted for T1 (baselines) in the primary working memory outcomes of visuo-spatial working memory (VSWM), visual working memory (VWM), and executive function (EF) as measured by the neuropsychological tests (Rey Auditory Test, Wechsler Adult Intelligence Scale [WAIS] IV symbol test, WAIS IV coding test, Delis-Kaplan Executive Function System [DKFES] color tests, Trails A and Trails B tests, and WAIS IV Letter and Number sequencing test) and self-report Patient Reported Outcomes Measurement Information System (PROMIS) surveys (Applied Cognition General Concerns Short Form, Applied Cognition Executive Function Short Form, and Functional Assessment of Cancer Therapy [FACT] Cognitive Function) between the intervention group and wait control group.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I (COMPUTER-ASSISTED COGNITIVE TRAINING): Patients complete a computerized working memory training program (Cogmed) over 35 minutes a day, 5 times a week for 6 weeks.

ARM II (WAIT LIST): Patients undergo standard follow-up care for 6 weeks. Following standard follow-up care, patients may complete Cogmed as in the Intervention Group in weeks 7-13.

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer (stage 0, I, II, III), 18 months to 5 years post oncologic therapies of surgery, chemotherapy, and/or radiation therapy (does not exclude current selective estrogen receptor modulators or aromatase inhibitors)
* Able to read, write, and speak English
* Mini Mental State Exam score greater than or equal to 19
* Have reliable internet and daily access to computer with audio/speakers
* Agree to travel to the Seattle Cancer Care Alliance (SCCA) or University of Washington (UW) School of Nursing for 2-3 in person assessments over the 12-13 weeks of the study

Exclusion Criteria:

* History of multiple cancers
* History of central nervous system (CNS) disease, CNS radiation, intrathecal therapy, or CNS surgery
* History of traumatic brain injury
* Neurologic disorders of stroke, encephalitis, dementia, epilepsy, Alzheimer's disease, Parkinson's disease
* Self-report of learning disabilities
* Substance addiction
* Diagnosis of psychiatric disorders of psychosis, schizophrenia, or bipolar disorder
* Mini mental state exam score less than 19
* Previous participation in cognitive training program
* Visual impairments such as uncorrected vision or color blindness
* Uncorrected hearing impairments
* Self-report that they are not pregnant or planning to become pregnant in the next four months
* Anticipate moving from the region in the next 4 months
* Inability to use a mouse or computer keys to navigate around the computer screen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-05; Primary Completion 2016-12-13 (Actual); Study Completion 2017-11-30 (Actual)

PRIMARY OUTCOMES:
Attrition rate | Up to 7 weeks
  Intervention completion percentage rate and the maximum level achieved for each working memory cognitive domain will be determined for each participant.
Percentage of participants retained in the study | Up to 7 weeks
  Intervention completion percentage rate and the maximum level achieved for each working memory cognitive domain will be determined for each participant.
Percentage of participants who are recruited | Up to 7 weeks
  Intervention completion percentage rate and the maximum level achieved for each working memory cognitive domain will be determined for each participant.
Satisfaction, measured by the satisfaction survey | Up to 7 weeks
  Satisfaction is measured on a 7-point Likert item questionnaire. The frequencies and the mode will be estimated from the satisfaction survey.

SECONDARY OUTCOMES:
Anxiety | Baseline to up to 7 weeks
  PROMIS Emotional Distress-Anxiety-Short Form.
Cognition | Baseline to up to 7 weeks
  FACT Cognitive Function, PROMIS Applied Cognition General Concerns Short Form, and Applied Cognition Executive Function Short Form.
Depression | Baseline to up to 7 weeks
  PROMIS Emotional Distress -Depression Short Form.
Executive Function | Baseline to up to 7 weeks
  D-KEFS color word tests, Trails A and B, and Letter-number sequencing.
Fatigue | Baseline to up to 7 weeks
  PROMIS Fatigue-Short Form.
Verbal Working Memory | Baseline to up to 7 weeks
  REY auditory verbal word memory recall and recognition test.
Visuo Spatial Working Memory | Baseline to up to 7 weeks
  Symbol recognition and coding test.

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Shannon Dorcy, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States